CLINICAL TRIAL: NCT04345939
Title: Rapid and Accurate Detection of Major Mycobacterium Species in Pulmonary
Brief Title: Rapid and Accurate Detection of Major Mycobacterium Species in Pulmonary Infection Based on GenSeizer Platform
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Haiqng Chu, Director, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: L20-203Y
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Mycobacterium Pulmonary Infection
MeSH Terms: interventions — Ovulation Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GenSeizer: Sputum and lavage fluids are tested for pathogens using GenSeizer
  Interventions: Diagnostic Test: Detection method
- PCR reverse hybridization: Sputum and lavage fluids are tested for pathogens using PCR reverse hybridization
  Interventions: Diagnostic Test: Detection method
- Target sequencing after incubation: Sputum and lavage fluids are tested for pathogens using Target sequencing after incubation
  Interventions: Diagnostic Test: Detection method

INTERVENTIONS:
Diagnostic Test: Detection method — Different methods for pathogen diagnosis

SUMMARY:
Comparison of rapid detection methods of mycobacterial pathogens, GenSeizer v.s. PCR reverse hybridization.

DETAILED DESCRIPTION:
The investigators developed a new platform called GenSeizer, which combines bioinformatics analysis of a large dataset with multiplex PCR-based targeted gene sequencing, to identify eleven major Mycobacterium species implicated in human disease. Simultaneous detection of certain antibiotic resistance genotypes, i.e., erm(41) and rrl in M. abscessus, is also feasible. This platform detected both reference strains and clinical isolates with a high degree of specificity and sensitivity.

In this study, the investigators plan to verify the detection efficiency of GenSeizer in clinical samples (sputum, alveolar lavage fluid) and compare it with existing methods on the market (PCR reverse hybridization) and gold standard method (target sequencing after incubation)

ELIGIBILITY:
Inclusion Criteria:

* Suspected cases of mycobacterial lung infection

Exclusion Criteria:

* No sputum
* Refused or unable to tolerate bronchoscopy

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Suspected cases of mycobacterial lung infection
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Detection accuracy | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Haiqing Chu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No